CLINICAL TRIAL: NCT02611583
Title: Double-blind, Randomized, Placebo Controlled Trial of Transcutaneous Electrical Nerve Stimulation (TENS) Treatment Plus Ibuprofen for the Treatment of Acute Back Pain in the Emergency Department
Brief Title: TENS Treatment Plus Ibuprofen for the Treatment of Acute Back Pain in the ED
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Never initiated due to lack of funding and IRB Approval
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Principal Investigator, Paul Dominici, MD, Albert Einstein Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HN4810
Record Dates: First submitted 2015-11-19; First posted 2015-11-23 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-03

CONDITIONS: Low Back Pain
Keywords: TENS
MeSH Terms: conditions — Low Back Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ibuprofen and TENS plus (Active Comparator): Patients will receive 45 minutes of TENS therapy. All patients will receive ibuprofen.
  Interventions: Device: TENS
- Ibuprofen and Sham TENS plus (Placebo Comparator): Patients will receive 45 minutes of sham TENS therapy. All patients will receive ibuprofen.
  Interventions: Device: TENS

INTERVENTIONS:
Device: TENS — Transcutaneous Electrical Nerve Stimulation

SUMMARY:
Patients presenting to the ED with a chief complaint of acute low back pain and whom the providing physician feels symptomatic treatment is appropriate in the ED will be screened for inclusion in the study. The purpose of the study is to compare Transcutaneous Electrical Nerve Stimulation (TENS) as an adjunct to ibuprofen in the treatment of acute low back pain in the emergency department. Therefore, the aim of this prospective, randomized, double blind study is to evaluate the efficacy of ED administered TENS in acute low back pain patients during their ED visit.

DETAILED DESCRIPTION:
The study is a double blind, randomized, placebo controlled trial. One group will receive ibuprofen and TENS. The comparison group will receive ibuprofen and sham TENS. The study primary endpoint is change in pain level on Visual Analog Scale score at 45-60 minutes after TENS start.

This is a two-arm, double blind, randomized control trial evaluating the patient perceived improvement in back pain. Patients will first fill out a Visual Analog Scale (VAS).

Patients will be randomized to one of two arms. Ibuprofen 800 mg, plus sham TENS for 45 minutes Ibuprofen 800 mg, plus TENS for 45 minutes

Patients will be given a 2nd VAS scale up to 15 minutes after the end of the TENS session. After the second VAS the patients will be finished with the study procedures and can be continued to be cared as per the discretion of their treating physician.

Our intention is to detect a 20% reduction in pain by VAS with a common standard deviation equal to the difference at the p = 0.05 level with a power of 80% using an analysis of variance (ANOVA). The calculated sample size required 28 patients per group. Considering the uncertain dropout rate, the investigators decided to enroll at least 66 patients. Baseline characteristics will be calculated to determine if groups are equal. A two-way repeated-measures ANOVA will be used to test both a trial effect and a group effect (SPSS 20, SPSS Inc., Chicago, IL). Data will be presented as means with standard deviations with 95% confidence intervals. A p< 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years to 65 years of age presenting to the emergency room with a primary complaint of low back pain.
2. Patient is receiving 800mg dose of ibuprofen as part of their treatment regimen for back pain
3. Back pain new in the last 48 hours
4. Deemed by the treating physician to have musculoskeletal back pain, and no central/peripheral nervous system pathology as the cause of their pain.

Exclusion Criteria:

1. Allergy to ibuprofen.
2. Hypotension (MAP <65 or Systolic BP <100), fever, tachycardia
3. Paresthesias, isolated motor weakness, or objective sensory deficit on physical exam
4. Radicular symptoms
5. Urinary incontinence or retention
6. Bowel incontinence
7. Unexplained weight loss of >15 lbs in the last 3 months.
8. Multiple primary complaints in the ED.
9. Received Analgesia other than Ibuprofen as part of their ED work up.
10. Taken prescription strength pain medication within the last 12 hours for any condition.
11. History of active malignancy, HIV, organ transplantation, active hemodialysis
12. Currently pregnant
13. Nursing home residents
14. Currently in police custody

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06-24 (Actual); Primary Completion 2016-06-24 (Actual); Study Completion 2016-06-24 (Actual)

PRIMARY OUTCOMES:
Change in visual analog scale (VAS) | 0 minutes, 45 minutes
  Patients will have a baseline and 45 minutes VAS performed

SECONDARY OUTCOMES:
Treatment failure | 45 minutes
  Patients requiring rescue medication after 45 minute treatment will be considered treatment failures and will receive further non study related treatment at the discretion of the treating physician
Adverse events | 60 minutes
  Any reactions to TENS application

CONTACTS AND LOCATIONS:
Overall Officials: Paul G Dominici, MD, Principal Investigator — Albert Einstein Healthcare Network
Locations (1):
- Albert Einstein Healthcare Network, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Cypress BK. Characteristics of physician visits for back symptoms: a national perspective. Am J Public Health. 1983 Apr;73(4):389-95. doi: 10.2105/ajph.73.4.389. PMID 6219588
- [Background] Patrick N, Emanski E, Knaub MA. Acute and chronic low back pain. Med Clin North Am. 2014 Jul;98(4):777-89, xii. doi: 10.1016/j.mcna.2014.03.005. PMID 24994051
- [Background] Thorsteinsson G, Stonnington HH, Stillwell KG, Elveback LR. The placebo effect of transcutaneous electrical stimulation. Pain. 1978 Jun;5(1):31-41. doi: 10.1016/0304-3959(78)90022-2. PMID 353652
- [Background] Marchand S, Charest J, Li J, Chenard JR, Lavignolle B, Laurencelle L. Is TENS purely a placebo effect? A controlled study on chronic low back pain. Pain. 1993 Jul;54(1):99-106. doi: 10.1016/0304-3959(93)90104-W. PMID 8378107
- [Background] Bertalanffy A, Kober A, Bertalanffy P, Gustorff B, Gore O, Adel S, Hoerauf K. Transcutaneous electrical nerve stimulation reduces acute low back pain during emergency transport. Acad Emerg Med. 2005 Jul;12(7):607-11. doi: 10.1197/j.aem.2005.01.013. PMID 15995091